CLINICAL TRIAL: NCT03410511
Title: Reversibility of Propylene Glycol/Glycerol Intake Effects on Cardiorespiratory Function
Brief Title: Propylene Glycol/Glycerol Intake and Cardiorespiratory Function
Acronym: PGGICF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Martin Chaumont, Principal investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P2016/466 / B406201629930
Record Dates: First submitted 2018-01-11; First posted 2018-01-25 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotine free intake (Experimental): The participant will wean off nicotine during five days before the experimental session. At the start of the experimental session, participants will be exposed to acute propylene glycol/glycerol (mix 50:50) intake.
  Interventions: Other: Nicotine free intake
- Nicotine intake (Experimental): The participant will pursuit his regular nicotinic propylene/glycerol intake five days before the experimental session. At the start of the experimental session, participants will be exposed to acute propylene glycol/glycerol/nicotine (mix 50:50) intake.
  Interventions: Other: Nicotine intake
- Cessation intake (Experimental): The participant will completely stop his regular nicotinic propylene/glycerol intake during five days before the session. At the start of the experimental session, participants will mimick intake with the device turns off.
  Interventions: Other: Cessation intake

INTERVENTIONS:
Other: Nicotine free intake — The participant will wean off nicotine during five days before the experimental session. At the start of the experimental session, participants will be exposed to acute propylene glycol/glycerol (mix 50:50) intake.
  Arms: Nicotine free intake
Other: Nicotine intake — The participant will pursuit his regular nicotinic propylene/glycerol intake five days before the experimental session. At the start of the experimental session, participants will be exposed to acute propylene glycol/glycerol (mix 50:50) intake.
  Arms: Nicotine intake
Other: Cessation intake — The participant will completely stop his regular nicotinic propylene/glycerol intake during five days before the session. At the start of the experimental session, participants will mimick intake with the device turns off.
  Arms: Cessation intake

SUMMARY:
Propylene glycol/Glycerol intake is increasingly popular. The propylene glycol/glycerol intake effects on cardiorespiratory function are unknown.

DETAILED DESCRIPTION:
Background. Propylene glycol/Glycerol intake is increasingly popular. The propylene glycol/glycerol intake effects on cardiorespiratory function are unknown. Weaning of propylene glycol/glycerol could allows a quick clearance of propylene glycol/glycerol from the body, with subsequent recovery of cardiorespiratory function.

Specific aim of the research. This research proposal tests the following hypothesis regarding the reversibility of propylene glycol/glycerol and nicotine intake:

* Propylene glycol/glycerol cessation restores cardiorespiratory function.
* Chronic propylene glycol/glycerol and propylene glycol/glycerol/nicotine intake induces specific serum and urine proteomics profile, which are partially reversed after cessation.
* Chronic propylene glycol/glycerol and propylene glycol/glycerol/nicotine intake induces specific serum and urine metabolomics profile, which are partially reversed after cessation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be regular propylene glycol/glycerol/nicotine intake users since at least 1 year
* Subject must be former smokers

Exclusion Criteria:

* Chronic or acute illness
* Substance abuse
* Chronic medication intake

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory function | 4 hours
  Continuous monitoring of cardiorespiratory function

SECONDARY OUTCOMES:
Change in serum and urine proteomics profiles | 1 hour
  Serum and urine proteomics

OTHER OUTCOMES:
Change in serum and exhaled breath condensate metabolomics profiles | 1 hour
  Serum and exhaled breath condensate metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Philippe van de Borne, MD, PhD, Study Director — Université Libre de Bruxelles
Locations (1):
- Erasme Hospital, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Any purpose Proposals should be directed to martin.chaumont@ulb.ac.be

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03410511/Prot_SAP_ICF_000.pdf